CLINICAL TRIAL: NCT03948152
Title: A Study to Determine Clinician and Patient Preferences Towards Interface Products Recommended by the 3D Mask Advice Tool
Brief Title: A Study to Determine Preferences Towards Interface Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SRC-SLE(PI)-CP-2018-10129
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Sleep Disorder; Breathing-Related
Keywords: Sleep Apnea
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea Syndromes | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care
- Mask Advice Tool (Experimental)
  Interventions: Other: Mask Advice Tool

INTERVENTIONS:
Other: Standard of Care — Participants will have a Positive Airway Pressure (PAP) mask chosen to wear for a period of 90 days as provided by the sites standard of care.
  Arms: Standard of Care
Other: Mask Advice Tool — Participants will have a Positive Airway Pressure (PAP) mask chosen to wear for a period of 90 days as provided by the mask advice tool.
  Arms: Mask Advice Tool

SUMMARY:
Enrolled Naïve participants will be randomized to one of two arms, the investigational or control arm. Once randomized the institutions will fit the participant with the procedures outlined in the protocol. Each participant will be required to trial the mask for a period of 90 days. Any Unscheduled Visits or Calls that occur during the participants 90 days documented.

ELIGIBILITY:
Inclusion Criteria:

* Adult Volunteers (ages 21-85)
* Willing and able to provide informed consent
* Able to follow instructions
* Able to read and speak in English as their primary language
* Currently diagnosed with Sleep Apnea through an in-lab sleep (polysomnography (PSG)) or home sleep testing, but has not started therapy and/or been fit with a mask.

Exclusion Criteria:

* Pre-existing conditions such as bullous lung disease, pathologically low blood pressure, bypassed upper airway, pneumothorax, pneumocephalus, cerebral spinal fluid (CSF) leaks, cribriform plate abnormalities, and prior history of head trauma that has resulted in current cognitive dysfunction.
* Prescribed an Adaptive Servo Ventilation (ASV) device
* The presence of physical or mental limitations that would limit the ability to test the mask.
* Obstructive Sleep Apnea (OSA) diagnosis achieved through a split night sleep study
* Known allergy to silicone
* Unique facial features (i.e. deformities of the face and/or head, piercings, etc) that could interfere with the use of masks.
* Employee of Philips or spouse of a Philips employee
* Currently participating in another interventional research study or planned participation in another interventional research study during the trial period (by self-report)
* Surgery involving the eyes, ears, nose, sinuses, or upper airway within the last 90 days.
* Planned surgical procedures involving the head, neck, face (eyes, ears, nose), or lung during the trial period.
* Uncontrolled or poorly managed gastroesophageal reflux
* Impaired cough reflex
* Untreated or symptomatic hiatal hernia
* Untreated glaucoma
* Untreated chronic dry eyes
* Unable to remove the sleep apnea mask without the assistance of others
* Use of prescription drugs that induce vomiting

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants requiring one or more mask re-fits | 90 days
  Proportion of participants in each arm requiring one or more mask re-fits.

SECONDARY OUTCOMES:
Number of masks tried during the initial fitting visit | 90 days
  Number of masks tried during the initial fitting visit in each arm.
Number of masks tried after going home with the first mask | 90 days
  Number of masks tried after going home with the first mask in each arm.
Amount of time to fit each mask | 90 days
  Amount of time to fit each mask in each arm.
Number of sleep clinic or sleep center callbacks related to mask fitting issues | 90 days
  Number of sleep clinic or sleep center callbacks related to mask fitting issues in each arm.
The amount of time spent on these calls to resolve mask issues | 90 days
  The amount of time spent on these calls to resolve mask issues in each arm.
Number of unplanned visits to adjust current mask or fit with another masks | 90 days
  Number of unplanned visits to adjust current mask or fit with another masks in each arm.
Duration of the unplanned visits | 90 days
  Duration of the unplanned visits in each arm.
Adherence to CPAP therapy | 90 days
  Adherence to CPAP therapy as determined by average hours of use
Mask leak for chosen masks | 90 days
  Mask leak for chosen masks in each arm.
Subjective preference rated by patients | 90 days
  Patients will complete a "Post-Trial Questionnaire" to rate their post-trial experience, on a 0-10 scale. "0" meaning strongly disagree/unlikely, "10" meaning strongly agree/likely. A higher score means a better outcome.
Subjective preference rated by clinicians | 90 days
  Clinicians will complete a "Post-Trial Questionnaire" to rate their post-trial experience, on a 0-10 scale. "0" meaning strongly disagree/unlikely, "10" meaning strongly agree/likely. A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pulmonary Disease Specialists, PA, d/b/a PDS Research, Kissimmee, Florida
  - Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Pullmonary Rehabilition Associates, Youngstown, Ohio
  - Berks Schuylkill Respiratory Specialists, Ltd., Reading, Pennsylvania
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No